CLINICAL TRIAL: NCT04643210
Title: The Management of My Bipolarity Intervention on the Combined Use of Technology and Face to Face Education on the Empowerment of Ill Health Self-management Skills in Adults With a Bipolar Disorder
Brief Title: Management of my Bipolarity Intervention in Bipolar Disorder Patients
Acronym: MoB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cyprus University of Technology (Other)
Responsible Party: Principal Investigator, Maria Karanikola, Accosiate Professor, Cyprus University of Technology
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5.34.01.7.6Ε/0490/2018; EEBK/EΠ/2018/27 (Other: CYPRUS NATIONAL BIOETHICS COMMITTEE)
Record Dates: First submitted 2020-10-21; First posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Bipolar Disorder; Affective Psychosis, Bipolar; Manic-Depressive Psychosis; Depression, Bipolar
Keywords: Education; Empowerment; Bipolar Disorder; Self-management
MeSH Terms: conditions — Bipolar Disorder; Empowerment

STUDY DESIGN:
Intervention Model Description: The study is a combination of a qualitative and a quantitative, interventional (quasi experimental) design. A focus group and content analysis will be implemented for the qualitative assessment of the educational needs of adults with a bipolar disorder. The educational intervention (MoB EI) will be developed according to the qualitative data on patients' educational needs and relevant literature, aiming to include combination of face to face (F2F) and technology-based interventions via design of a Digital platform. The effectiveness of the MoB EI regarding the acquired self-management skill will be assessed via structured instruments in the quantitative part of the study using descriptive and inferential statistics (SPSS version 24.0).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- F2F MoB EI and access to MoB Digital Platform (MoB DP) group (Experimental): The design of the face-to-face Management of my Bipolarity educational intervention (F2F MoB EI) will rely on the Colom & Vieta model, Cognitive- Behavioural techniques and the results of the relevant literature review and data acquired in the qualitative research of bipolar disease patients' educational needs. A textbook will be devised explaining in detail the step-by-step process and the techniques of the experimental educational method of the MoB F2F EI.
  This group will also receive the technology-based intervetion, which regards access to the MoB DP. This is an ecosystem where the participants will be educated and empowered making use of the internet of things (IOT) via a computer, tablet or mobile.
  Interventions: Behavioral: F2F MoB EI; Other: MoB DP
- The MoB DP group (Active Comparator): This group will receive the technology-based intervention, which regards access to the MoB DP. The structure of the MoB DP has been partially based on the preferences and needs of the participants (as described in the qualitative part of the study) and its goal is to create an ecosystem where users will be educated and empowered making use of the internet of things (IOT) via a computer, tablet or mobile. The Digital platform will be in the form of a dynamic website with user generated content as well as static information.
  Interventions: Other: MoB DP

INTERVENTIONS:
Behavioral: F2F MoB EI — The MoB F2F EI will comprise a total of 12 educational F2F sessions. Each session will have a duration of 1.5 hours and the maximum number of participants in the groups will be 12 patients.
  The intervention group will receive the MoB F2F EI on group or personal form according to the participant's choice. The implementation methodology of the MoB F2F EI will include videos and power point presentations, as well as interactive learning methods such as role-playing, empowerment exercises, live discussions.
  Arms: F2F MoB EI and access to MoB Digital Platform (MoB DP) group
Other: MoB DP — This is a technology-based intervention, which regards access to a dfigital platform, the MoB DP. The structure of the Digital platform has been partially based on the preferences and needs of the participants (as described in the qualitative part of the study) and its goal is to create an ecosystem where users will be educated and empowered making use of the internet of things (IOT) via a computer, tablet or mobile. The Digital platform will be in the form of a dynamic website with user generated content as well as static information.

SUMMARY:
The Management of my Bipolarity study aims to develop an educational intervention (MoB EI) on the combined use of technology and face to face education on the empowerment of ill health self-management skills in adults with bipolar disorder. The MoB EI will be developed according to qualitative data on patients' educational needs and relevant literature. The effectiveness of acquired knowledge and self-management skills will be assessed according to the degree of a) cognitive functioning, b) impulse control, c) adherence to pharmacotherapy, d) relapse prevention, d) improvement of quality of life of participants.

DETAILED DESCRIPTION:
The aim of the study is to develop and test an educational intervention for patients with bipolar disorder (BD). The objectives include:

1. A literature review on BD educational programs.
2. Exploration of the educational needs of adults with BD.
3. Development of the MoB educational intervention (MoB EI), encompassing a face to face (F2F) intervention and a technology-based intervention via a Digital platform (MoB DP).
4. Exploration of the effectiveness of the MoB EI in BD patients regarding i) their knowledge on BD, and ii) empowerment of ill health self-management skills in relation to the improvement of impulse control, adherence to pharmacotherapy, relapse frequency, quality of life and adaptive attitudes towards substance use.

Design This study uses a mixed-method design and consists of four stages.

Stage 1: (a) To conduct a literature review on BD educational programs, and (b) define the educational needs of adults with BD via empirical exploration of their living experience (a focus group and content analysis will be implemented for this qualitative assessment), aiming to integrate both data in the MoB EI.

Stage 2: Design of the MoB F2F EI & the MoB Digital Platform (MoB DP). ΜoΒ F2F EI:The design of this intervention will rely on the Colom & Vieta model, Cognitive- Behavioural techniques and the results of the 1st stage (all relevant literature and data acquired in the qualitative research of educational needs). A textbook will be devised explaining in detail the step-by-step process and the techniques of the experimental educational method of the MoB F2F EI.

MoB DP: The structure of the MoB DP has been designed by the researchers of the present study and a web developer, partially based on the preferences and needs of the participants (as described in Stage 1); its goal is to create an ecosystem where people with BD will be educated and empowered making use of the internet of things (IOT) via a computer, tablet or mobile. The MoB DP will be in the form of a dynamic website with user generated content as well as static information. A responsive design has been applied, i.e. accessible by all types of devices. The platform is accessible to the participants in the current study, as well as to any interested person, e.g., family members of people with BP, or care givers providing updated information related to BD (platform users). The platform administrator is the main researcher (AH), while the owner is the Nursing Department of the Cyprus University of Technology (CUT). The participants of the proposed study will have the opportunity to access the platform both during and after the completion of the study.

The informative part of the platform is live (www.mob.com.cy), while the interactive part is under development. The informative part, so far, includes the following functionalities: self-management action plan, home-work exercises, self-assessment tools, scientific articles relevant to BD. Entry into the platform functionalities (scientific articles excluded) is password protected.

Specifically, the users of the platform will have the opportunity to register by filling in their personal profile and revisit when they wish. Regarding self-management functionalities, the platform will contain subject units where personal relapse symptoms may be registered, a life events table, personal risk factors for relapse and a weekly program of activities. Input of relevant information will be through open-ended questions and check lists. Participants of the MoB F2F EI who visit the platform, will find that these subject units (chapters) are topics on which they will be educated on. Additional features will be incorporated according to development of 1st stage, e.g., new training needs, as described by participants in the focus groups.

Another subject unit will be the personal therapy file, where users will have the chance to keep tabulated notes related to their therapy, including information about the dose and type of medication treatment, as well as pending medical test, e.g., blood test, and other relevant information. The therapeutic team of the user will have the possibility to register in the platform under the approval of the user with the aim to support continuity and sharing of information.

Stage 3: Implementation and evaluation of the effectiveness of the MoB EI. All eligible participants will be assigned into the intervention group and the control group. Based on power analysis the intervention group will be constituted of 40 participants and the control (waiting) group of 40 participants.

The criteria for discontinuing participation in intervention group are disorder relapse and non-adherence to pharmacotherapy (discontinuation of medication).

Intervention description. The intervention group will receive the MoB F2F EI on group or personal form according to the participant's choice. Also the participants of the intervention group will have access to the MoB DP.

The implementation methodology of the MoB F2F EI will include videos and power point presentations, as well as interactive learning methods such as role-playing, empowerment exercises, live discussions.

The MoB F2F EI will comprise a total of 12 educational F2F sessions. Each session will have a duration of 1.5 hours and the maximum number of participants in the groups will be 12 patients. At the beginning of each session, the participants will be given the opportunity to record their feedback for the previous session and the impact of the training program, so far, on them and their families / significant others. The location where the MoB F2F EI will be conducted is the CUT. The main researcher (AH) will implement the MoB F2F EI. Participation in the educational intervention is free of charge. Also, no economic outcomes are expected to emerge through this or any stage of the study.

Those who will wish to withdraw before completion of the intervention, will be able to continue to receive information/knowledge about their illness through the digital platform.

The control group will have access only to the MoB DP.

Effectiveness evaluation. The evaluation of the effectiveness of the MoB F2F EI will be based on the degree of improvement on the following parameters:

1. Self-perceived quality of life level
2. Ability to control impulses
3. Psychoactive substances use attitudes
4. Adherence to pharmacotherapy
5. Frequency of relapses
6. BD Knowledge level

There will be four evaluation timepoints. The 1st evaluation timepoint will be prior to the implementation of the MoB F2F EI, the 2nd will take place immediately after the completion of the MoB F2F EI, while the 3rd and 4th ones will be applied six and twelve months, respectively, after the completion of the MoB EI. These timepoints have been determined according to relevant literature.

The control group will be assessed via the same evaluation tools as the intervention group, and at the same time periods.

This will verify the hypothesis that patients who receive only pharmacotherapy and have access to the MoB DP do not have the same improvement as intervention group in important aspects of their lives, i.e., quality of life, cognitive functioning, impulse control, adherence to pharmacotherapy, relapse prevention.

Data analysis. Mean and standard deviation will be assessed for the scale numeric scores (WHOQOL, DUDIT, MoCa, DAI-30, relapse frequency) and frequencies will be tested for categorical variables (gender, age groups, group years in illness). Parametric tests (ANOVA, t-test) will be applied for comparisons between groups. For all statistical tests, p values of 0.05 or lower will be considered statistically significant. Data will be analysed through the Statistical Package for Social Sciences (SPSS, Inc, Chicago, IL version 25.00). To test the relationship between two or more variables logistic and linear regression analysis will be used. Regarding missing data, multiple imputation method will be applied.

Stage 4: Assessment of the applicability of the Digital platform. The assessment of the applicability of the digital platform will be based on qualitative (users' feedback) and quantitative testing (data analysis). Regarding users' qualitative feedback, there will be an exploration of the experience of the users with the platform and the degree to which they were positively affected by its use. This process will take place via focus groups discussions. The focus of the interviews will be on the impact of the platform on their everyday life, as well as on enhancement of ill health self-management skills. It is intended to deliver 2 focus groups with 8-12 participants each. The participants will be among those who (a) attended the F2F EI and at the same time had used the platform, (b) only had access to the MoB DP.

The evaluation of the platform will also take place through anonymous questionnaires by asking the users of the platform to answer predefined questions regarding satisfaction parameters relevant to the platform. The technology which will be applied for this process is Google Forms. This part of the assessment is expected to take place during the second half of 2021.

ELIGIBILITY:
Inclusion criteria:

1. Clinical diagnosis based on DSM-5 for BD type I and II.
2. Age between 18 and 65.
3. Signed informed consent.
4. Stabilized mood status at the beginning of the MoB F2F intervention based on clinical assessment, conducted by the primary investigator (AH).
5. Experience of the illness of at least one year based on reported medical record.
6. Adequate awareness of the illness, based on the following guide: (a) are you aware of the reason(s) you are using mental health services/ under medication? and (b) are you aware of the aim of the educational intervention in which you may participate?

Exclusion criteria:

1. Intellectual disability (IQ<70), based on the Wechsler Adult Intelligence Scale (WAIS).
2. Brain damage (e.g, following a stroke), based on diagnostic tests.
3. Acute phase of the illness which requires hospitalization.
4. Acute phase of the illness, based on clinical assessment, as well as the Young Mania Rating Scale (YMRS) and/or Beck's Depression Inventory (BDI) tools.
5. Substance use problems at the beginning of this stage according to the Alcohol Use Disorders Identification Test (AUDIT) and Drug Use Disorders Identification Test (DUDIT) tools.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Bipolar disease patients educational needs | 6 months
  Qualitative measures: 1. Knowledge/ mental health literacy on present medical condition (measurement tool [MT]/ Open-ended question: Please tell us, what do you know about your mental health condition/ BD?) 2. Knowledge gap regarding BD (MT/ Open ended question: Please describe what you would like to know about bipolar disorders).
  3. Topics to be covered (MT/ Open ended question: Please describe in what way/topics you would like to be educated on bipolar disorders/to increase your knowledge about bipolar disorders? 4. Educational and feasibility expectations (MT/ Open-ended questions: a. Please describe your expectations from an educational program regarding the impact on your everyday living b. How you would like this program to be implemented one on one or in a group? C. How long would you like the program to last? 5. e-Health literacy (MT/ Open ended question: What is your level of engagement with the Internet?)
Degree of self-perceived quality of life as measured by the total score in the scale "World Health Organization Quality of Life Assessment". | 18 months
  The scale "World Health Organization Quality of Life Assessment" is a 1-5 Likert type scale including 26 items. The minimum score in the scale is 26 and the maximun is 130.
  Higher scores indicate a better outcome.
Level of knowledge regarding BD, as measured by the total score in the scale "Bipolar Disorder Knowledge Scale". | 18 months
  The "Bipolar Disorder Knowledge Scale" is a 25-item true-false scale. The scale assesses knowledge of BD with items targeting diagnosis, etiology, disease course, symptoms, treatment, and life impact. The ration of "true" to "false" responses is assessed. Higher percentage values indicate a better outcome.
Degree of ability to control impulses, as measured by the total score in the scale "YOUNG MANIA RATING SCALE " (YMRS) . | 18 months
  The "YMRS" is a 0-4 likert scale, including 11 items. The total score of the scale ranges from 0 to 44. The lower the total score the better the outcome.
Degree of adherence to pharmacotherapy, as measured by the total score in the scale "Drug Attitude Inventory" (DAI). | 18 months
  The "DAI" is a 30 item "true-false" scale.The ration of "true" to "false" responses is assessed. Higher percentage values indicate a better outcome.
Degree of dysfunctional attitudes towards substance use as measured by the total score in the scale "Drug Use Disorders Identification Test" (DUDIT). | 18 months
  The scale DUDIT is a 1-5 Likert, 11-item scale (scale total score range: 1-55) . The lower the total score the better the outcome.
  Lower scores indicate a better outcome.
Degree of dysfunctional attitudes towards alcohol as measured by the total score in the scale "Alcohol Use Disorders Identification Test" (AUDIT). | 18 months
  The AUDIT scale is a 0-4 Likert, 10-item scale (scale total score range: 0-40) .
  Lower scores indicate a better outcome.
Frequency of relapses, as measured by the number of hospitalizations after the completion of the face to face intervention. | Two years following the end of the face tot face educational intervention.
  The number of hospitalizations will be measured as the sum of the individual hospitalizations in a high security psychaitric hospital.
  The lower the number of the frequency the better the outcome.
Reduced duration of relapses, as measured by the duration of inpatient hospitalizations in days after the completion of the face to face intervention. | Two years following the end of the face to face educational intervention.
  The duration of inpatient hospitalizations will be measured as the sum of the days of hospitalization in high security psychaitric hospitals.
  The lower the duration in days of the hospitalization the better the outcome.
Degree of feasibility of the digital platform, as measured by users' qualitative feedback on the following open-ended question: "Please tell us, what was your experience with the MoB DP use? | 6 months
  The more positive the described experience the better the outcome.
Degree of feasibility of the digital platform, as measured by the users' qualitative feedback on the impact of the MoB DP on their life based on the following open-ended question: "Please tell us, what was the impact of the MoB DP use on your life?" | 6 months
  The more positive the described impact of the MoB DP on users' life the better the outcome.
Degree of feasibility of the digital platform, measured by users' feedback on the impact of the platform on their self-management skills based on the question "What was the impact of the platform on your ill health self-management skills?" | 6 months
  The more positive the described impact of the digital platform on users' ill health self-management skills the better the outcome.
Degree of feasibility of the digital platform, as measured by users' self-reported degree of satisfaction on MoB DP by the total score on the scale "Users' Satisfaction Scale" (USS). | 6 months
  The USS is 1-3 Likert scale (low;moderate/accepted; high), which includes 6 items, assessing users' perceptions about overall experienced satisfaction (item1); utility according to their present medical condition (item 2); feasibility on daily usage (item 3); technical difficulties experienced (item 4); improvement of BD self-management skills (item 5); improvement of BD knowledge (item 6).
  The total score of the USS ranges between 6- 18. The higher the total score the better the outcome.

SECONDARY OUTCOMES:
Description of the topics of the MoB educational intervention through a qualitative measure. | 6 months
  Measurement tool: Open-ended question "Please describe on which topics you would like to be aducated or increase your knowledge on BD with focus on therapeutic issues, pathophysiology, well-being and patients' rights."
Description of the mode of the MoB educational intervention through a qualitative measure. | 6 months
  Measurement tool: Open-ended question "Please describe the mode through which you would like to recieve information with special focus on the duration, number of sessions and duration of each session of the intervention"
Description of the different modes of the MoB educational intervention through a qualitative measure. | 6 months
  Measurement tool: Open-ended question "Please describe the mode through which you would like to recieve information with focus on personal or group sessions, face-to-face or via internet sessions "
Description of the MoB DP technology-based intervention through a qualitative measure. | 6 months
  Measurement tool: Open-ended question "What is your preferences regarding a technology-based educational intervention on BD with focus on the topics to be included, on the information provision mode (interactive or not), and access modes (tablet, mobile, personal computer)?"

CONTACTS AND LOCATIONS:
Overall Officials: Maria NK Karanikola, Study Chair — Cyprus University of Technology
Locations (1):
- Cyprus University of Technology, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Through publications
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: After the end of the study and for the next 5 years
Access Criteria: These will be decided upon the end of the study

REFERENCES:
- [Background] 21. Hatzioannou A, Papastavrou E, Chatzittofis A, Karanikola M. Exploration of the effectiveness of structured education in empowering people with Bipolar Disorder. Nursing Care & Research 2020;55:246-274.
- [Derived] Hatzioannou A, Chatzittofis A, Koutroubas VS, Papastavrou E, Karanikola M. Combined Use of Web-Based and In-Person Education on Ill Health Self-management Skills in Adults With Bipolar Disorder: Protocol for a Mixed Methods Study. JMIR Res Protoc. 2021 Sep 8;10(9):e25168. doi: 10.2196/25168. PMID 34494969